CLINICAL TRIAL: NCT06161896
Title: Characterization and Clinical Impact of the Gut Microbiota in Diffuse Large B-cell Lymphoma Patients
Brief Title: Characterization and Clinical Impact of the Gut Microbiota in Lymphoma
Status: Recruiting | Type: Observational
Sponsor: Lars Møller Pedersen (Other)
Collaborators: Zealand University Hospital (Other); Herlev Hospital (Other); Statens Serum Institut (Other); Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor-Investigator, Lars Møller Pedersen, MD, PhD, Herlev Hospital
Organization: Herlev Hospital (Other)
Other Study IDs: MiCheLin
Record Dates: First submitted 2023-11-15; First posted 2023-12-08 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fecal and blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DLBCL cohort: Interventions for the DLBCL cohort are:
  * Fecal samples
  * Blood samples
  * Bioelectrical impedance analyses
  * Filling in questionnaires
  All other procedures will be in accordance with local and national guidelines corresponding to clinical standard care.
  Interventions: Diagnostic Test: Stool samples
- Healthy control cohort: The control group applied in the current study is based on the Danish General Suburban Population Study (GESUS). The control subjects are selected from the GESUS cohort and matched according to age and gender.
  Serial stool samples are planned in a subset of the control cohort with sampling time points corresponding to the DLBCL cohort. The sample material is handled and stored the same way as for the DLBCL cohort.
  Interventions: Diagnostic Test: Stool samples

INTERVENTIONS:
Diagnostic Test: Stool samples — Analysis of microbiome, mutations, alterations in body composition and lifestyle
  Other Names: Blood samples; Bioelectrical impedance analysis; Questionnaires

SUMMARY:
The study is a prospective observational single-center cohort study which compare the gut microbiome of newly diagnosed Diffuse Large B-cell Lymphoma patients with the gut microbiome of healthy controls. Furthermore the impact of lymphoma treatment, immune phenotypes, cytokine profiles, metabolomics, inflammation, driver mutations, comorbidity, body composition and lifestyle on the microbiome is also investigated

DETAILED DESCRIPTION:
Microbiota refers to an ecological community of commensal, symbiotic and pathogenic microorganisms that colonize the various compartments within the human body including the gastrointestinal tract. The composition has been shown to play an important role in the pathophysiology of many diseases as well as influence host homeostatic processes such as regulation of metabolic processes, defense against pathogens, immune system development, regulation of the immune response and inflammation. However, the connection between the gut microbiota and lymphoma remain poorly understood.

The purpose of this study is to evaluate the composition and diversity of the gut microbiome in a large homogeneous group of patients with newly diagnosed and treatment-naive Diffuse Large B-cell Lymphoma (DLBCL). The investigators aim to identify the relationship between the intestinal microbiota, clinical and molecular subtypes of DLBCL and outcome of the disease. The association between nutrition, physical activity, body composition, toxicity to the antineoplastic therapy, infections, use of antibiotics, comorbidity and tumor genetics versus gut microbiota composition and diversity is also explored.

The project is carried out in collaboration between clinical departments, institutes and laboratories with expertise in microbiology, hematology, pathology, nutrition, molecular biology, immunology and bioinformatics.

Hypothesis of the study are:

1. Patients with DLBCL have distinct baseline microbiota signatures that differ from healthy subjects.
2. Significant changes in the microbiota composition and diversity can be identified during and after treatment (immunochemotherapy) of DLBCL.
3. Lymphoma response and outcome is affected by the composition and diversity of the DLBCL microbiota.
4. The intestinal microbiota changes towards a microbiota more like the microbiota of healthy controls in patients who remain in lymphoma remission one year after completion of therapy.
5. Distinct DLBCL microbiota profiles are associated with treatment-related toxicity.
6. The intestinal microbiota affects the risk of infections (clinically and/or microbiologically documented).
7. The intestinal microbiota is affected using antibiotics both as prophylaxis and treatment of infections.
8. The DLBCL microbiota depends on the dietary intake, smoking, physical activity and the body composition.
9. Distinct intestinal microbiota signatures can be associated with molecular subtypes of DLBCL (or vice versa)
10. The JAK2V617F, TET2, DNMT3A and ASXL1 mutations affect the intestinal microbiota signature and are associated with comorbidity and outcome in DLBCL
11. There is a vicious circle between intestinal dysbiosis and lymphoma with the crosstalk between the gut microbiota and the cancer being expressed as alterations in the profile of cytokines, chemokines and growth factors; an immune response reflected by immunophenotypic profiles of peripheral blood mononuclear cells; and characteristic metabolite signatures in the blood.

ELIGIBILITY:
Inclusion Criteria for the DLBCL cohort:

* WHO 2022 classified newly diagnosed and treatment-naïve large B-cell lymphoma (DLBCL) belonging to one of the following entities:
* Diffuse large B-cell lymphoma, including transformation from an indolent lymphoma
* Follicular lymphoma grade 3B
* T-cell/histiocyte-rich LBCL
* Primary cutaneous DLBCL, leg type
* EBV-positive DLBCL, NOS
* Primary mediastinal LBCL
* High grade B-cell lymphoma with MYC/BCL2 rearrangement
* The patient is a candidate for R-CHOP-like first-line treatment
* Staging by PET available before treatment initiation
* Age ≥18 years
* Written informed consent

Exclusion Criteria for the DLBCL cohort:

* Pregnancy
* Psychiatric illness or condition which could interfere with their ability to understand the requirements of the study
* Clinical signs of uncontrolled serious infection
* Clinical gastrointestinal lymphoma involvement
* Other significant gastrointestinal comorbidities
* Any other prior malignancy than non-melanoma skin cancer or stage 0 (in situ), cervical carcinoma, unless treated with curative intent, and without relapse for 2 years, or low-grade prostate cancer, not in need of treatment
* Ileostomy
* CNS involvement at diagnosis
* Severe cardiac disease: NYHA grade 3-4
* Impaired liver (transaminases > 3 x normal upper limit or bilirubin > 1.5 x normal upper limit, unless due to Gilbert´s syndrome) or renal (GFR<30ml/min) function not caused by lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include two different cohorts:
  A: Newly diagnosed and treatment-naïve DLBCL patients
  B: A healthy control cohort
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Intestinal microbiota baseline characterization | 1.5 years
  Assessment using amplicon-based sequencing of ribosomal (r)RNA genes

SECONDARY OUTCOMES:
Intestinal microbiota characterization at mid-, post-treatment and at follow up | 2.5 years
  Assessment using amplicon-based sequencing of ribosomal (r)RNA genes
Assessment of habitual diet | 2.5 years
  Food frequency questionnaire (FFQ)
Assessment of energy and macronutrient intake | 2.5 years
  24h dietary recalls
Assessment of physical activity | 2.5 years
  International physical activity questionnaire (IPAQ)
Body composition | 2.5 years
  Body composition according to bioelectrical impedance analysis (BIA) using BioScan touch i8 - IVF version
Smoking | 2.5 years
  Packages (baseline lifestyle questionnaire)
Alcohol intake | 2.5 years
  Units (baseline lifestyle questionnaire)
Treatment-related toxicity | 1.5 years
  Treatment-related toxicity (CTCAE criteria)
Antibiotics | 1.5 years
  Use of any type of prophylactic and therapeutic antibiotics during treatment (baseline lifestyle questionnaire)
Statins | 1.5 years
  Use of any type of statins during treatment registered in the Shared Medication Record (FMK)
Medication | 1.5 years
  Use of any type of medication registered in the Shared Medication Record (FMK)
Infections | 1.5 years
  Clinical infections during treatment
Lymphoma response | 1.5 years
  Lymphoma response after completion of first line treatment (Lugano criteria)
Molecular signatures | 1.5 years
  Molecular signatures in standard clinical practice according to Hans classification (cell of origin (COO))
Chromosome abnormalities | 1.5 years
  Molecular signatures in standard clinical practice (fluorescent in situ hybridization (FISH))
Mutations | 1.5 years
  JAK2V617F, TET2, DNMT3A and ASXL1 mutation analyses (%VAF)
Cytokine profiles | 1.5 years
  Magnetic bead-based assays
Metabolite signatures | 1.5 years
  Metabolomic profiling by a combination of GC and LC coupled with MS
Peripheral blood mononuclear cell (PBMC) profiles | 1.5 years
  PBMC profiles according to flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Sophie Staxen, MSc, Principal Investigator — Zealand University Hospital - Roskilde
Locations (1):
- Zealand University Hospital, Department of Hematology, Roskilde, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.